CLINICAL TRIAL: NCT01957033
Title: Clinical and Biological Responses of People With Neck Pain Being Treated With Varying Doses of Manual Therapy: A Pilot Study
Brief Title: Responses of People With Neck Pain Being Treated With Varying Doses of Manual Therapy: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan Miller, Graduate Student (Other)
Collaborators: Physiotherapy Foundation of Canada (Unknown)
Responsible Party: Sponsor-Investigator, Jordan Miller, Graduate Student, Graduate student, School of Rehabilitation Science, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 13-569
Record Dates: First submitted 2013-09-29; First posted 2013-10-08 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Whiplash Injuries
Keywords: whiplash; neck pain; manual therapy; exercise; dosage
MeSH Terms: conditions — Whiplash Injuries; Neck Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (9):
- Duration 6 weeks, frequency 3/week (Experimental): Exercise and education 3 times/week for 6 weeks Manual therapy 3 times/week for 6 weeks
  Interventions: Behavioral: Exercise and education 3 times/week for 6 weeks; Other: Manual therapy 3 times/week for 6 weeks
- Duration 6 weeks, Frequency twice/week (Experimental): Exercise and education twice/week for 6 weeks Manual therapy twice/week for 6 weeks
  Interventions: Behavioral: Exercise and education twice/week for 6 weeks; Other: Manual therapy twice/week for 6 weeks
- Duration 6 weeks, Frequency once/week (Experimental): Exercise and education once/week for 6 weeks Manual therapy once/week for first 6 weeks
  Interventions: Behavioral: Exercise and education once/week for 6 weeks; Other: Manual therapy once/week for 6 weeks
- Duration 3 weeks, Frequency 3 times/week (Experimental): Exercise and education 3 times/week for 6 weeks Manual therapy 3 times/week for first 3 weeks
  Interventions: Behavioral: Exercise and education 3 times/week for 6 weeks; Other: Manual therapy 3 times/week for 3 weeks
- Duration 3 weeks, Frequency twice/week (Experimental): Exercise and education twice/week for 6 weeks Manual therapy twice/week for first 3 weeks
  Interventions: Behavioral: Exercise and education twice/week for 6 weeks; Other: Manual therapy twice/week for 3 weeks
- Duration 3 weeks, frequency once/week (Experimental): Exercise and education once/week for 6 weeks Manual therapy once/week for first 3 weeks
  Interventions: Behavioral: Exercise and education once/week for 6 weeks; Other: Manual therapy once/week for 3 weeks
- Duration 0 weeks, Frequency 3 times/week (Experimental): Exercise and education 3 times/week for 6 weeks No manual therapy
  Interventions: Behavioral: Exercise and education 3 times/week for 6 weeks
- Duration 0 weeks, Frequency twice/week (Experimental): Exercise and education twice/week for 6 weeks. No manual therapy
  Interventions: Behavioral: Exercise and education twice/week for 6 weeks
- Duration 0 weeks, Frequency once/week (Experimental): Exercise and education once/week for 6 weeks No manual therapy
  Interventions: Behavioral: Exercise and education once/week for 6 weeks

INTERVENTIONS:
Behavioral: Exercise and education once/week for 6 weeks — Exercises will include specific range of motion, strengthening, and motor control exercises for the neck and shoulder girdle. Education will include prognosis information, advice to stay active, and use of a book
  Arms: Duration 0 weeks, Frequency once/week; Duration 3 weeks, frequency once/week; Duration 6 weeks, Frequency once/week
Behavioral: Exercise and education twice/week for 6 weeks — Exercises will include specific range of motion, strengthening, and motor control exercises for the neck and shoulder girdle. Education will include prognosis information, advice to stay active, and use of a book about whiplash.
  Arms: Duration 0 weeks, Frequency twice/week; Duration 3 weeks, Frequency twice/week; Duration 6 weeks, Frequency twice/week
Behavioral: Exercise and education 3 times/week for 6 weeks — Exercises will include specific range of motion, strengthening, and motor control exercises for the neck and shoulder girdle. Education will include prognosis information, advice to stay active, and use of a book about whiplash.
  Arms: Duration 0 weeks, Frequency 3 times/week; Duration 3 weeks, Frequency 3 times/week; Duration 6 weeks, frequency 3/week
Other: Manual therapy once/week for 3 weeks — Manual therapy will consist of low velocity mobilizations of the cervical and upper thoracic spine based on the findings of the treating physiotherapist.
  Arms: Duration 3 weeks, frequency once/week
Other: Manual therapy twice/week for 3 weeks — Manual therapy will consist of low velocity mobilizations of the cervical and upper thoracic spine based on the findings of the treating physiotherapist.
  Arms: Duration 3 weeks, Frequency twice/week
Other: Manual therapy 3 times/week for 3 weeks — Manual therapy will consist of low velocity mobilizations of the cervical and upper thoracic spine based on the findings of the treating physiotherapist.
  Arms: Duration 3 weeks, Frequency 3 times/week
Other: Manual therapy once/week for 6 weeks — Manual therapy will consist of low velocity mobilizations of the cervical and upper thoracic spine based on the findings of the treating physiotherapist.
  Arms: Duration 6 weeks, Frequency once/week
Other: Manual therapy twice/week for 6 weeks — Manual therapy will consist of low velocity mobilizations of the cervical and upper thoracic spine based on the findings of the treating physiotherapist.
  Arms: Duration 6 weeks, Frequency twice/week
Other: Manual therapy 3 times/week for 6 weeks — Manual therapy will consist of low velocity mobilizations of the cervical and upper thoracic spine based on the findings of the treating physiotherapist.
  Arms: Duration 6 weeks, frequency 3/week

SUMMARY:
The purpose of this pilot project is to determine the feasibility of a study design to investigate how many sessions of manual therapy and exercise produce the best results for people with whiplash injuries. Also, this study will help us determine the best way to measure the effect of treatment. Finally, the investigators will study how closely the physiotherapists follow the treatment instruction provided in the study protocol and training. In order to achieve these objectives, 12 people will receive manual therapy and exercise at one of twelve different doses. the investigators will have each of these people fill out questionnaires, measure sensation changes, and measure changes in the way people move their necks while walking. This study will help us determine if the study protocol can be carried out as planned. This includes: the training of all people involved in carrying out the assessments and treatments, the willingness and ability of participants to take part in all of the treatment and measures involved. This will provide us with important information to help us plan a larger study with 226 people with whiplash injuries.

ELIGIBILITY:
Inclusion Criteria:

* adults ≥ 21 years
* main complaint must be neck pain, but we expect some patients will also report symptoms that radiate to the shoulder and arm regions or have an associated headache.
* pain intensity must be ≥ 12/40 on the 4-item pain scale (P4).

Exclusion Criteria:

* non-mechanical sources of neck pain or over-riding comorbidity listed below:
* rheumatoid arthritis
* neurological diseases
* fractures
* dislocation
* rheumatoid arthritis
* upper motor neuron dysfunction or malignancy
* pregnant women
* closed head injury
* on steroid-based medications within the past 6 months.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-10; Primary Completion 2015-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Feasibility | 1 year
  As a pilot study, the main outcome of interest is feasibility. This includes: ability to train assessors and health care providers, time it takes to complete all assessments, ability to recruit 12 patients within 1 year, and completeness of data collected.
Pain | 12 weeks (end of treatment) and 6- and 12- month follow-ups
  Measured by the 4-item pain questionnaire (P4). This will be a primary outcome of the full trial.
Function | 12 weeks (end of treatment) and 6- and 12- month follow-up
  Measured by the Neck Disability Index (NDI). This will be a primary outcome measure of the full powered study.

SECONDARY OUTCOMES:
Fidelity | 1 year
  As a pilot study, the secondary outcome of interest is treatment fidelity. We will measure this through ability of health care providers to provide treatment at the dosage described in the protocol.
Psychological measures | 12 weeks (end of treatment)
  Catastrophic thinking measured by Pain Catastrophizing Scale (PCS) Anxiety and Depression measured by Hospital Anxiety and Depression Scale (HADS) Psychological distress measured by Trauma Anxiety and Distress Scale (TADS)
Psychophysical measures | 12 weeks (end of treatment)
  Vibration Pain Threshold (VPT), Current Perception Threshold (CPT), Pressure Pain Threshold (PPT), Response to Cold Provocation(RCP)
Motor coordination | 12 weeks (end of treatment)
  Neck Walk Index (NWI)
Health Status | 12 weeks (end of study) and 6- and 12- month follow-ups
  Measured by SF-36
Global perceived effect | 12 weeks (end of treatment) and 6- and 12-month follow-ups
  Global perceived effect will be measured on a 7 point scale (-3 to +3)
Upper extremity function | 12 weeks (end of treatment) and 6- and 12-month follow-ups
  As measured by the shortened version of the Disability of the Arm, Shoulder, Hand (qDASH).

CONTACTS AND LOCATIONS:
Overall Officials: Jordan D Miller, MSc, Principal Investigator — McMaster University; Joy C MacDermid, PhD, Principal Investigator — McMaster University
Locations (3):
- Canada (3):
  - McMaster Univervisty, Hamilton, Ontario
  - Lifemark Health, Hamilton, Hamilton, Ontario
  - Western University, London, Ontario